CLINICAL TRIAL: NCT04918303
Title: Skin Sympathetic Nerve Activity and Cardiac Arrhythmia
Acronym: SKNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2020/55
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Sudden Death; Ventricular Tachycardia; Persistent Atrial Fibrillation
Keywords: Skin sympathetic nerve activity (SKNA); Electrocardiogram (ECG); Cardiac arrythmia
MeSH Terms: conditions — Death, Sudden; Tachycardia, Ventricular; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SKNA group (Experimental)
  Interventions: Device: SKNA recording

INTERVENTIONS:
Device: SKNA recording — The coupled recording of the sympathetic nervous activity of the skin and of an ECG will be carried out using the ME6000 device, CE marked, from the Bittium company.
  It will be performed for a maximum period of one hour at Day 1, Post-procedure between Day 1 and discharge from hospital, and month 6

SUMMARY:
Sympathetic tone is important in cardiac arrhythmogenesis. The simultaneous recording of sympathetic nerve activity (SNA) and electrocardiogram (ECG) was obtained by invasive method. The purpose of this protocol is to further develop this recording method to turn it into a new non-invasive tool for arrhythmia prediction and detection. This method may also be useful in validating the results of surgical procedures aimed at sympathetic denervation

ELIGIBILITY:
Inclusion Criteria:

- patient hospitalized at Bordeaux University Hospital for sudden death, ventricular tachycardia, persistent or paroxysmal atrial fibrillation treated by ablation and/or vein of Marshall ethanol infusion

Exclusion Criteria:

* pregnancy,
* patient under 18 year old,
* patient with a cardiac stimulation device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Delay between the discharge of the sympathetic system and the rhythmic event. | Day 1
  Temporal correlation of occurrence of sympathetic electrical event and cardiac arrhythmia by the MacNemar test will be performed.
Delay between the discharge of the sympathetic system and the rhythmic event. | Day 2
  Temporal correlation of occurrence of sympathetic electrical event and cardiac arrhythmia by the MacNemar test will be performed.
Delay between the discharge of the sympathetic system and the rhythmic event. | Month 6
  Temporal correlation of occurrence of sympathetic electrical event and cardiac arrhythmia by the MacNemar test will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Mélèze Hocini, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France